CLINICAL TRIAL: NCT02853032
Title: Image-guided, Robotically Delivered Transcranial Magnetic Stimulation Treatment for Combat-Related Post-Traumatic Stress Disorder: a Double-Blind, Randomized Comparison to Sham Transcranial Magnetic Stimulation
Brief Title: Image-guided, Robotically Delivered Transcranial Magnetic Stimulation Treatment for Combat-Related Post-Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Laurel Ridge Treatment Center (Other); Consortium to Alleviate PTSD (Other)
Responsible Party: Principal Investigator, Felipe S. Salinas, Ph.D., Assistant Professor--Research, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC20160191H
Record Dates: First submitted 2016-07-25; First posted 2016-08-02 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active rTMS to the right DLPFC (Active Comparator): Active repetitive transcranial magnetic stimulation will be delivered to the right DLPFC using connectivity-based, image-guided aiming with the rTMS coil positioned using a robotic arm. In this arm, active rTMS will be delivered at 20 Hertz (Hz) in 2 sec trains with 14 sec inter-train intervals, 20 minutes/session (i.e. 1,600 pulses/session), 7 days/week for 20 consecutive days.
  Interventions: Device: Active repetitive transcranial magnetic stimulation; Device: robotic arm
- Sham rTMS to the right DLPFC (Placebo Comparator): Sham repetitive transcranial magnetic stimulation will be delivered to the right DLPFC using connectivity-based, image-guided aiming with the rTMS coil positioned using a robotic arm. In this arm, sham rTMS will be delivered at 20 Hz in 2 sec trains with 14 sec inter-train intervals, 20 minutes/session (i.e. 1,600 pulses/session), 7 days/week for 20 consecutive days.
  Interventions: Device: robotic arm; Device: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Active repetitive transcranial magnetic stimulation — The MagPro R30 is an advanced, high performance magnetic stimulator designed primarily for non-invasive clinical use. The non-invasive brain stimulation system will be used to deliver active repetitive electromagnetic pulses in this research study's treatment of post-traumatic stress disorder.
  Other Names: rTMS
  Arms: Active rTMS to the right DLPFC
Device: robotic arm — This robotic system is based on a commercially available neurosurgical robot. The robot is mounted on a mobile (i.e. retractable wheels) cart which holds the robot controller and the TMS power supply and pulse-generation computer. The robotic system will be used for TMS coil positioning/targeting.
Device: Sham repetitive transcranial magnetic stimulation — The MagPro R30 is an advanced, high performance magnetic stimulator designed primarily for non-invasive clinical use. The non-invasive brain stimulation system will be used to deliver placebo repetitive electromagnetic pulses in this research study's treatment of post-traumatic stress disorder.
  Other Names: sham rTMS
  Arms: Sham rTMS to the right DLPFC

SUMMARY:
Mounting amounts of evidence suggests that non-invasive stimulation of the dorsolateral prefrontal cortex (DLPFC) using repetitive transcranial magnetic stimulation (rTMS) maybe a safe and effective treatment modality for Post-Traumatic Stress Disorder (PTSD). However the large variability in the magnitude of clinical outcomes reported is likely related to the current lack of knowledge of ideal side of stimulation (left vs right) and the limited precision in the targeting of brain circuits needed to obtain an optimal treatment response. In this protocol the investigators will: 1) generate individualized treatment plans based on an individual's functional Magnetic Resonance Imaging (fMRI) and meta-analytical based connectivity analysis to guide the delivery of adjunct, imaging-based & robotically delivered rTMS to active duty military (ADM) subjects with PTSD participating in an intensive program providing integrated evidence-based psychotherapy and pharmacological management (Treatment as Usual (TAU)). 2) To use clinician ratings and self-report PTSD symptom scales, as well as other indicators of clinical change, to determine whether compared with TAU, addition of adjunct rTMS improves clinical outcomes. 3) To conduct neuroimaging-based assessments aimed to measure rTMS effects on network connectivity in ADM receiving treatment for PTSD and the potential correlation of connectivity changes with clinical outcomes.

DETAILED DESCRIPTION:
The investigators propose a randomized, double-blind, sham-controlled, 20 consecutive day trial of adjunct rTMS to the right DLPFC for ADM with PTSD receiving TAU at Laurel Ridge Treatment Center (LRTC; San Antonio, TX). Methods: Consenting ADM receiving TAU for PTSD at LRTC will be randomized to receive 20 consecutive days of adjunct rTMS according to one of these two treatment arms: Arm 1 TAU plus rTMS to the right DLPFC and Arm 2 TAU plus sham rTMS. At UTHSCSA's Research Imaging Institute (RII), where all brain imaging will be conducted, rTMS treatment plans will be generated based on (pre-treatment) anatomical and functional magnetic resonance imaging (fMRI) to guide the optimal robotic positioning of the TMS coil to accurately target each subject's DLPFC. Initial diagnostic interview and weekly clinical follows ups will be conducted at the LRTC by research clinicians blinded to subjects' research group. A comparison of baseline brain connectivity measurements with subjects' neuroimaging follow ups conducted at treatment Week 3 will be conducted to identify network connectivity changes potentially associated to treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female English-speaking active duty or recently retired veteran patients who have deployed post 9/11 receiving treatment at LRTC between the ages of 18-65 years;
2. Patients must have a diagnosis of PTSD confirmed by the Clinician-Administered PTSD Scale (CAPS-5) at screening,
3. Subjects must have a minimum PTSD Symptom Checklist (PCL-5) for DSM-V symptom severity rating of 25.

Exclusion Criteria:

1. Subjects with a diagnostic history of bipolar disorder, schizophrenia or schizoaffective disorder as documented in the medical record.
2. Substance use disorder during the 12 months prior to screening; except that Mild - Moderate, but not Severe, Alcohol Use Disorder (using DSM-5 criteria) will be allowed as determined by LRTC medical provider review.
3. Any history or signs of serious medical or neurological illness including seizure disorders. Except for seizures, a subject with a clinical abnormality may be included only if the study clinician considers the illness will not introduce additional risk and will not interfere with the study procedures. This will be determined during the screening phase via self-report and/or medical history review.
4. History of traumatic brain injury (TBI) with loss of consciousness for 20 minutes or more as determined by the History of Head Injuries questionnaire.
5. Females will be excluded if they are pregnant (i.e. positive pregnancy test identified after their LRTC intake).
6. Any history or signs of metal objects deemed unsafe for MRI or that may adversely affect image quality of the brain region (e.g. surgical clips, cardiac pacemakers, metal implants, etc.) in the body at the time of screening as indicated by self-report. MRI can have risks for persons with foreign bodies implanted in their body.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe S Salinas, Ph.D., Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Laurel Ridge Treatment Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data at this time.

REFERENCES:
- [Result] Boggio PS, Rocha M, Oliveira MO, Fecteau S, Cohen RB, Campanha C, Ferreira-Santos E, Meleiro A, Corchs F, Zaghi S, Pascual-Leone A, Fregni F. Noninvasive brain stimulation with high-frequency and low-intensity repetitive transcranial magnetic stimulation treatment for posttraumatic stress disorder. J Clin Psychiatry. 2010 Aug;71(8):992-9. doi: 10.4088/JCP.08m04638blu. Epub 2009 Dec 29. PMID 20051219

RESULTS

PARTICIPANT FLOW:
Groups:
- Active rTMS to Right DLPFC: Active repetitive transcranial magnetic stimulation will be delivered to the right DLPFC using connectivity-based, image-guided aiming with the rTMS coil positioned using a robotic arm.
- Sham rTMS to the Right DLPFC: Sham repetitive transcranial magnetic stimulation will be delivered to the right DLPFC using connectivity-based, image-guided aiming with the rTMS coil positioned using a robotic arm.
Period: Overall Study
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Started | 60 | 59
Completed | 51 ("Evaluable" = 10 or more irTMS sessions "Completers" = 15 or more irTMS sessions) | 56 ("Evaluable" = 10 or more irTMS sessions "Completers" = 15 or more irTMS sessions)
Not Completed | 9 | 3
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Requested to withdraw from all treatment | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.48 (7.02) | 38.60 (6.35) | 38.10 (6.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 55 | 52 | 107
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 12 | 14 | 26
  White | 40 | 39 | 79
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 59 | 119

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Severity as Measured by the PTSD Checklist (PCL-5)
Description: The PCL-5 is a 20-item measure that assesses the presence and severity of PTSD symptoms. Responders are asked to rate how bothered they have been by each item in the past month on a 5-point Likert scale ranging from 0-4. Items are summed to provide a total score. Severity can be determined adding scores of each item together to determine a total score. The range is 0-80, with a lower score suggesting a lower incidence of PTSD. A total score of 33 or higher suggests the patient needs further assessment to confirm a diagnosis of PTSD.
Time Frame: Baseline to three weeks (the conclusion of rTMS treatment)
Population: Discrepancies in the number of participants analyzed for this outcome measure occur because of 1) incomplete assessments at the designated outcome measure's time frame or 2) because the participant did not complete more than 15 treatment sessions, but were considered "evaluable" (>10 sessions).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 55 | 58
score on a scale
  baseline | 59.82 (10.07) | 60.45 (11.74)
  3 weeks: number analyzed (Participants) | 51 | 58
  3 weeks | 33.29 (19.86) | 39.14 (19.35)

2. Secondary Outcome: Change in Depression Severity as Measured by the 9-item Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 is a brief, 9-item scale that includes only the depression-related items from the PHQ. The PHQ-9 has been validated for use in primary care settings and can be used to make a tentative diagnosis of depression and to monitor depression severity and response to treatment in the past 2 weeks. Higher scores indicate increasing depressive symptoms. Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe. Remission from severe depression is defined as a PHQ-9 score less than or equal to 14.
Time Frame: Baseline to three weeks (the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active rTMS to the Right DLPFC: Active repetitive transcranial magnetic stimulation will be delivered to the right DLPFC using connectivity-based, image-guided aiming with the rTMS coil positioned using a robotic arm. In this arm, active rTMS will be delivered at 20 Hertz (Hz) in 2 sec trains with 28 sec inter-train intervals, 20 minutes/session (i.e. 1,600 pulses/session), 7 days/week; 20 consecutive days.
  Active repetitive transcranial magnetic stimulation: The MagPro R30 is an advanced, high performance magnetic stimulator designed primarily for non-invasive clinical use. The non-invasive brain stimulation system will be used to deliver active repetitive electromagnetic pulses in this research study's treatment of post-traumatic stress disorder.
  robotic arm: This robotic system is based on a commercially available neurosurgical robot. The robot is mounted on a mobile (i.e. retractable wheels) cart which holds the robot controller and the TMS power supply and pulse-generation computer. The robotic system w
- Sham rTMS to the Right DLPFC: Sham repetitive transcranial magnetic stimulation will be delivered to the right DLPFC using connectivity-based, image-guided aiming with the rTMS coil positioned using a robotic arm. In this arm, sham rTMS will be delivered at 20 Hz in 2 sec trains with 28 sec inter-train intervals, 20 minutes/session (i.e. 1,600 pulses/session), 7 days/week for 20 consecutive days.
  robotic arm: This robotic system is based on a commercially available neurosurgical robot. The robot is mounted on a mobile (i.e. retractable wheels) cart which holds the robot controller and the TMS power supply and pulse-generation computer. The robotic system will be used for TMS coil positioning/targeting.
  Sham repetitive transcranial magnetic stimulation: The MagPro R30 is an advanced, high performance magnetic stimulator designed primarily for non-invasive clinical use. The non-invasive brain stimulation system will be used to deliver placebo repetitive electromagnetic pulses in this research study's treatment
Arm/Group | Active rTMS to the Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 55 | 58
score on a scale
  baseline | 17.80 (5.24) | 19.31 (5.85)
  3 weeks: number analyzed (Participants) | 51 | 58
  3 weeks | 10.67 (6.73) | 12.19 (6.67)

3. Secondary Outcome: Change in Depression Severity as Measured by the Montgomery-Ashberg Depression Rating Scale (MADRS)
Description: The MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item yields a score of 0 to 6 and the overall score ranges from 0 to 60. Higher scores indicate increasing depressive symptoms. Cut-off points include: 0 to 6 - symptom absent, 7 to 19 - mild depression, 30 to 34 - moderate, 35 to 60 - severe depression.
Time Frame: Baseline to three weeks (the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS to the Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 55 | 58
score on a scale
  baseline | 25.55 (9.20) | 28.12 (9.28)
  3 weeks: number analyzed (Participants) | 51 | 58
  3 weeks | 13.96 (10.22) | 16.17 (10.31)

4. Secondary Outcome: Change in PTSD Severity as Measured by the PTSD Checklist for DSM-5 (PCL-5)
Description: as for outcome 1
Time Frame: Baseline to seven weeks (four weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 55 | 58
score on a scale
  baseline | 59.82 (10.07) | 60.45 (11.74)
  seven weeks: number analyzed (Participants) | 26 | 27
  seven weeks | 28.35 (14.57) | 40.22 (22.81)

5. Secondary Outcome: Change in PTSD Severity as Measured by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5)
Description: The CAPS-5 is a 30-item structured interview that can be used to make current (past month) diagnosis of PTSD, make lifetime diagnosis of PTSD, and assess PTSD symptoms over the past week. The assessor combines information about frequency and intensity of an item into a single severity rating. CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms; the range of the scores is 0-80; with a higher score indicating a higher incidence of PTSD symptoms. To meet criteria for PTSD, a patient must have:
  1. A traumatic event
  2. At least one "Re-experiencing" symptom
  3. At least one "Avoidance" symptom
  4. At least two "Negative alterations in cognitions and mood" symptoms
  5. At least two "Alterations in arousal and reactivity" symptoms
  6. The trauma must last at least a month
  7. The trauma must cause impairment
Time Frame: Baseline to seven weeks (four weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 55 | 58
score on a scale
  baseline | 45.05 (8.90) | 46.12 (8.14)
  seven weeks: number analyzed (Participants) | 24 | 20
  seven weeks | 24.83 (14.37) | 31.00 (12.86)

6. Secondary Outcome: Change in Depression Severity as Measured by the 9-item Patient Health Questionnaire (PHQ-9)
Description: as for outcome 2
Time Frame: Baseline to seven weeks (four weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 55 | 58
score on a scale
  baseline | 17.80 (5.24) | 19.31 (5.85)
  seven weeks: number analyzed (Participants) | 26 | 27
  seven weeks | 10.77 (6.21) | 14.19 (7.67)

7. Secondary Outcome: Change in Depression Severity as Measured by the Montgomery-Ashberg Depression Rating Scale (MADRS)
Description: as for outcome 3
Time Frame: Baseline to seven weeks (four weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 55 | 58
score on a scale
  baseline | 25.55 (9.20) | 28.12 (9.28)
  seven weeks: number analyzed (Participants) | 23 | 20
  seven weeks | 15.78 (11.74) | 19.75 (10.68)

8. Secondary Outcome: Change in PTSD Severity as Measured by the PTSD Checklist for DSM-5 (PCL-5)
Description: PCL-5 is a 20-item measure that assesses the presence and severity of PTSD symptoms. Responders are asked to rate how bothered they have been by each item in the past month on a 5-point Likert scale ranging from 0-4. Items are summed to provide a total score. Severity can be determined adding scores of each item together to determine a total score. The range is 0-80, with a lower score suggesting a lower incidence of PTSD. A total score of 33 or higher suggests the patient needs further assessment to confirm a diagnosis of PTSD.
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 55 | 58
score on a scale
  baseline | 59.82 (10.07) | 60.45 (11.74)
  sixteen weeks: number analyzed (Participants) | 15 | 14
  sixteen weeks | 34.47 (19.06) | 46.64 (22.61)

9. Secondary Outcome: Change in PTSD Severity as Measured by the Clinician-Administered PTSD Scale (CAPS-5)
Description: as for outcome 5
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 55 | 58
score on a scale
  baseline | 45.05 (8.90) | 46.12 (8.14)
  sixteen weeks: number analyzed (Participants) | 12 | 11
  sixteen weeks | 28.58 (14.27) | 31.45 (14.75)

10. Secondary Outcome: Change in Depression Severity as Measured by the 9-item Patient Health Questionnaire (PHQ-9)
Description: as for outcome 2
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 55 | 58
score on a scale
  baseline | 17.80 (5.24) | 19.31 (5.85)
  sixteen weeks: number analyzed (Participants) | 15 | 14
  sixteen weeks | 13.87 (7.31) | 16.86 (7.05)

11. Secondary Outcome: Change in Depression Severity as Measured by the Montgomery-Ashberg Depression Rating Scale (MADRS)
Description: as for outcome 3
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 55 | 58
score on a scale
  baseline | 25.55 (9.20) | 28.12 (9.28)
  16 weeks: number analyzed (Participants) | 12 | 12
  16 weeks | 20.50 (14.31) | 21.75 (12.54)

12. Secondary Outcome: Clinically Significant Response as Measured by the PTSD Checklist for DSM-5 (PCL-5)
Description: The PCL-5 is a 20-item measure that assesses the presence and severity of PTSD symptoms. Responders are asked to rate how bothered they have been by each item in the past month on a 5-point Likert scale ranging from 0-4. Items are summed to provide a total score. Severity can be determined adding scores of each item together to determine a total score. The range is 0-80, with a lower score suggesting a lower incidence of PTSD. A total score of 33 or higher suggests the patient needs further assessment to confirm a diagnosis of PTSD. A clinically significant response is defined as a 10-20 point decrease in the PCL-5 scores.
Time Frame: Baseline to three weeks (the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 51 | 58
percentage of change from baseline | -45.03 (4.47) | -36.53 (3.43)

13. Secondary Outcome: Clinically Significant Response in Depression Severity as Measured by the 9-item Patient Health Questionnaire (PHQ-9)
Description: as for outcome 2
Time Frame: Baseline to three weeks (the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 48 | 58
percentage of change from baseline | -37.04 (5.22) | -31.61 (5.86)

14. Secondary Outcome: Clinically Significant Response in Depression Severity as Measured by the Montgomery-Ashberg Depression Rating Scale (MADRS)
Description: The MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item yields a score of 0 to 6 and the overall score ranges from 0 to 60. Higher scores indicate increasing depressive symptoms. Cut-off points include: 0 to 6 - symptom absent, 7 to 19 - mild depression, 30 to 34 - moderate, 35 to 60 - severe depression. Clinically significant response is defined as greater than or equal to a 50% decrease in the MADRS score.
Time Frame: Baseline to three weeks (the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 49 | 58
percentage of change from baseline | -42.75 (5.29) | -40.74 (4.54)

15. Secondary Outcome: Clinically Significant Response as Measured by the PTSD Checklist for DSM-5 (PCL-5)
Description: as for outcome 12
Time Frame: Baseline to seven weeks (four weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 26 | 27
percentage of change from baseline | -50.44 (4.44) | -34.28 (5.86)

16. Secondary Outcome: Clinically Significant Response as Measured by the Clinician-Administered PTSD Scale (CAPS-5)
Description: The CAPS-5 is a 30-item structured interview that can be used to make current (past month) diagnosis of PTSD, make lifetime diagnosis of PTSD, and assess PTSD symptoms over the past week. The assessor combines information about frequency and intensity of an item into a single severity rating. CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms; the range of the scores is 0-80; with a higher score indicating a higher incidence of PTSD symptoms. To meet criteria for PTSD, a patient must have:
  1. A traumatic event
  2. At least one "Re-experiencing" symptom
  3. At least one "Avoidance" symptom
  4. At least two "Negative alterations in cognitions and mood" symptoms
  5. At least two "Alterations in arousal and reactivity" symptoms
  6. The trauma must last at least a month
  7. The trauma must cause impairment
  A clinically significant response is defined as at least a 50% decrease in the CAPS-5.
Time Frame: Baseline to seven weeks (four weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 24 | 20
percentage of change from baseline | -44.84 (5.52) | -29.59 (6.41)

17. Secondary Outcome: Clinically Significant Response in Depression Severity as Measured by the 9-item Patient Health Questionnaire (PHQ-9)
Description: as for outcome 2
Time Frame: Baseline to seven weeks (four weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 26 | 27
percentage of change from baseline | -34.47 (7.06) | -13.28 (11.51)

18. Secondary Outcome: Clinically Significant Response in Depression Severity as Measured by the Montgomery-Ashberg Depression Rating Scale (MADRS)
Description: as for outcome 14
Time Frame: Baseline to seven weeks (four weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 21 | 20
percentage of change from baseline | -23.40 (11.05) | -24.42 (10.30)

19. Secondary Outcome: Clinically Significant Response as Measured by the PTSD Checklist for DSM-5 (PCL-5)
Description: as for outcome 12
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 15 | 14
percentage of change from baseline | -40.20 (9.18) | -17.01 (9.80)

20. Secondary Outcome: Clinically Significant Response as Measured by the Clinician-Administered PTSD Scale (CAPS-5)
Description: as for outcome 16
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 12 | 11
percentage of change from baseline | -31.32 (13.00) | -27.64 (9.83)

21. Secondary Outcome: Clinically Significant Response in Depression Severity as Measured by the 9-item Patient Health Questionnaire (PHQ-9)
Description: as for outcome 2
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 15 | 14
percentage of change from baseline | -28.35 (11.18) | 19.36 (23.18)

22. Secondary Outcome: Clinically Significant Response in Depression Severity as Measured by the Montgomery-Ashberg Depression Rating Scale (MADRS)
Description: as for outcome 14
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 12 | 12
percentage of change from baseline | -22.65 (12.86) | -20.47 (12.34)

23. Secondary Outcome: Remission From PTSD as Measured by the PTSD Checklist for DSM-5 (PCL-5)
Description: The PCL-5 is a 20-item measure that assesses the presence and severity of PTSD symptoms. Responders are asked to rate how bothered they have been by each item in the past month on a 5-point Likert scale ranging from 0-4. Items are summed to provide a total score. Severity can be determined adding scores of each item together to determine a total score. The range is 0-80, with a lower score suggesting a lower incidence of PTSD. A total score of 33 or higher suggests the patient needs further assessment to confirm a diagnosis of PTSD. Remission is defined as a PCL-5 score less than or equal to 33.
Time Frame: Baseline to three weeks (the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of patients remitted
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 51 | 58
percentage of patients remitted | 58.82 | 46.55

24. Secondary Outcome: Remission From Depression as Measured by the 9-item Patient Health Questionnaire (PHQ-9)
Description: as for outcome 2
Time Frame: Baseline to three weeks (the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of patients remitted
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 48 | 58
percentage of patients remitted | 62.75 | 67.24

25. Secondary Outcome: Remission From Depression as Measured by the Montgomery-Ashberg Depression Rating Scale (MADRS)
Description: The MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item yields a score of 0 to 6 and the overall score ranges from 0 to 60. Higher scores indicate increasing depressive symptoms. Cut-off points include: 0 to 6 - symptom absent, 7 to 19 - mild depression, 30 to 34 - moderate, 35 to 60 - severe depression. Remission from depression is defined as a MADRS score less than or equal to 10.
Time Frame: Baseline to three weeks (the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of patients remitted
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 49 | 58
percentage of patients remitted | 45.10 | 39.66

26. Secondary Outcome: Remission From PTSD as Measured by the PTSD Checklist for DSM-5 (PCL-5)
Description: as for outcome 23
Time Frame: Baseline to seven weeks (four weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of patients remitted
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 26 | 27
percentage of patients remitted | 61.54 | 48.15

27. Secondary Outcome: Remission From PTSD as Measured by the Clinician-Administered PTSD Scale (CAPS-5)
Description: The CAPS-5 is a 30-item structured interview that can be used to make current (past month) diagnosis of PTSD, make lifetime diagnosis of PTSD, and assess PTSD symptoms over the past week. The assessor combines information about frequency and intensity of an item into a single severity rating. CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms; the range of the scores is 0-80; with a higher score indicating a higher incidence of PTSD symptoms. To meet criteria for PTSD, a patient must have:
  1. A traumatic event
  2. At least one "Re-experiencing" symptom
  3. At least one "Avoidance" symptom
  4. At least two "Negative alterations in cognitions and mood" symptoms
  5. At least two "Alterations in arousal and reactivity" symptoms
  6. The trauma must last at least a month
  7. The trauma must cause impairment
  Remission is defined as a CAPS-5 score less than or equal to 29.
Time Frame: Baseline to seven weeks (four weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of patients remitted
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 24 | 20
percentage of patients remitted | 54.17 | 45.00

28. Secondary Outcome: Remission From Depression as Measured by the 9-item Patient Health Questionnaire (PHQ-9)
Description: as for outcome 2
Time Frame: Baseline to seven weeks (four weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of patients remitted
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 26 | 27
percentage of patients remitted | 76.92 | 59.26

29. Secondary Outcome: Remission From Depression as Measured by the Montgomery-Ashberg Depression Rating Scale (MADRS)
Description: as for outcome 25
Time Frame: Baseline to seven weeks (four weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of patients remitted
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 21 | 20
percentage of patients remitted | 30.43 | 25.00

30. Secondary Outcome: Remission From PTSD as Measured by the PTSD Checklist for DSM-5 (PCL-5)
Description: as for outcome 23
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of patients remitted
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 15 | 14
percentage of patients remitted | 60.00 | 21.43

31. Secondary Outcome: Remission From PTSD as Measured by the Clinician-Administered PTSD Scale (CAPS-5)
Description: as for outcome 27
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of patients remitted
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 12 | 11
percentage of patients remitted | 41.67 | 27.27

32. Secondary Outcome: Remission From Depression as Measured by the 9-item Patient Health Questionnaire (PHQ-9)
Description: as for outcome 2
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of patients remitted
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 15 | 14
percentage of patients remitted | 60.00 | 35.71

33. Secondary Outcome: Remission From Depression as Measured by the Montgomery-Ashberg Depression Rating Scale (MADRS)
Description: as for outcome 25
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of patients remitted
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 12 | 12
percentage of patients remitted | 25.00 | 25.00

34. Secondary Outcome: Functional Connectivity Changes (Measured by Resting-state Functional Magnetic Resonance Imaging) of the Targeted Brain Network(s) Following rTMS Treatment
Description: Resting-state brain networks were identified using functional Magnetic Resonance Imaging. Any changes in the the targeted brain network (e.g. the sub-genual cingulate cortex) were reported using functional connectivity Z-scores. Functional connectivity Z-score indicates the number of standard deviations away from the baseline mean. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean, and lower connectivity, and positive numbers indicate values higher than the baseline mean, and higher connectivity
Time Frame: Baseline to three weeks (the conclusion of rTMS treatment)
Population: Functional brain connectivity to the sub-genual cingulate (SGC) cortex compared between the Active and Sham groups (in participants with >15 treatment sessions) at baseline and 3 weeks.
Measure: Number; unit: z-score
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 52 | 57
z-score | -1.02 | 1.17

35. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events and Serious Adverse Events
Description: This measure counts the number of participants with adverse events and serious adverse events.
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
Number analyzed (Participants) | 60 | 59
Participants
  AE | 36 | 32
  SAE | 0 | 0
  UPIRSO | 0 | 0
  none | 24 | 27

ADVERSE EVENTS:
Time Frame: Sixteen weeks
Arm/Group | Active rTMS to Right DLPFC | Sham rTMS to the Right DLPFC
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59
Other Adverse Events (participants affected / at risk) | 36/60 | 29/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active rTMS to Right DLPFC (N=60) | Sham rTMS to the Right DLPFC (N=59)
Headache (General disorders) | 16 | 19
Claustrophobia during MRI (General disorders) | 1 | 1
Increased Anxiety (General disorders) | 2 | 2
Numbness in Extremities (General disorders) | 1 | 0
Muscle Twitching (General disorders) | 5 | 1
Facial Discomfort (General disorders) | 6 | 0
Unable to tolerate TMS (General disorders) | 3 | 0
Vision Blurred (General disorders) | 1 | 0
Dizziness (General disorders) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT02853032/Prot_SAP_000.pdf